CLINICAL TRIAL: NCT01260740
Title: The Effect of Transcranial Magnetic Stimulation on Learning With Reward in Healthy Humans
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110055; 11-N-0055
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-06-23

CONDITIONS: Normal Physiology; fMRI
Keywords: Traumatic Brain Injury; Explicit Learning; Primary Motor Cortex; Dorsolateral Prefrontal Cortex; Implicit Learning; Healthy Volunteer; HV
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Two areas on the surface of the brain, the dorsolateral prefrontal cortex (DLPFC) and motor cortex (MC), play a key role during learning. Researchers are interested in determining the effect that transcranial magnetic stimulation (TMS) on the DLPFC and MC has on participants' performance of learning tasks. By studying the effect of TMS on reaction time, learning, and memory, researchers hope to better understand how to treat conditions such as Parkinson's disease and traumatic brain injury that affect these parts of the brain.

Objectives:

* To study the effects of transcranial magnetic stimulation on the dorsolateral prefrontal cortex and motor cortex.
* To learn which areas of the brain are used to perform certain learning and memory tasks.

Eligibility:

- Healthy, right-handed individuals between 18 and 70 years of age.

Design:

* Participants will be screened with a physical and neurological examination and a medical and psychiatric history.
* Participants will be asked to take part in one of five different parts of this study. Most participants will have four 2-hour visits to the National Institutes of Health Clinical Center. Some participants (those involved in Part 5) will have only one 2-hour visit.
* Parts 1 and 2 (four visits): Participants will have TMS, and then do a learning task that may provide a small monetary reward. On the first visit, before the TMS, participants will take an intelligence test based on reading aloud the words given on a card. Participants who have not had a routine magnetic resonance imaging (MRI) scan of the brain within the past year will also have a scan.
* Parts 3 and 4 (four visits): Participants will have a functional MRI scan while doing a learning task that may provide a small monetary reward. On the first visit, before the functional MRI, participants will take an intelligence test based on reading aloud the words given on a card. Participants who have not had a routine magnetic resonance imaging (MRI) scan of the brain within the past year will also have a scan.
* Part 5 (one visit): Participants will take an intelligence test based on reading aloud the words given on a card. Then, participants will have TMS followed by a functional MRI scan. During the functional MRI, participants will do a button-pressing task that may provide a small monetary reward.
* Participants will also be asked to provide a small blood sample for genetic analysis.

DETAILED DESCRIPTION:
Objective

Theta burst transcranial magnetic stimulation (TBS) produces functional changes in human motor cortex. Continuous inhibitory TBS, (cTBS) over the primary motor cortex (M1) produces a temporary impairment of learning in healthy individuals similar to that seen in patients with traumatic brain injury (TBI) and Parkinson disease (PD). The depression of learning by cTBS may serve as a model for learning and memory deficits in these disorders and provide a means of screening treatments for efficacy and exploring their mechanisms. Our immediate goal is to see whether manipulation of the behavioral contingencies of the task, particularly adding reward, will overcome the virtual lesion produced by cTBS.

The first aim of the project is to examine inhibitory effects of cTBS on implicit (serial reaction time /SRT) and explicit (trial-and-error) motor learning of a sequence of target locations.

The second aim of the project is to examine the effects of cTBS on non-motor implicit and explicit probabilistic classification learning using the weather prediction task (WPT). We will investigate the involvement of M1 and dorsolateral prefrontal cortex (DLPFC) in implicit and explicit learning by studying participants who will perform these tasks following cTBS over: 1) M1, 2) DLPFC and 3) sham TBS.

Our third aim is to examine the effect of manipulating reward during implicit and explicit learning following inhibitory TBS over M1 and DLPFC as it is possible that learning deficits caused by TBS can be improved by increasing the amount of reinforcement during learning.

Our fourth aim is to examine the neural networks underlying implicit and explicit learning with and without reward by studying participants who will perform these tasks during functional MRI (fMRI). Finally, we will also perform fMRI during implicit sequence learning and after cTBS over M1 to identify its effects on the neural networks involved in implicit learning.

Study population

Healthy volunteers (n = 272, aged 18 70), without any contraindication to TBS or MRI. This number includes 60 participants each for Experiments 1 and 2, 24 participants each for Experiments 3-5. In addition, 35 participants are included for piloting behavioral and imaging procedures. In order to account for potential dropouts and withdrawals (up to 20%), the total accrual ceiling includes a further 45 participants to equal 272.

Design

The study contains five, mixed or crossover design experiments with appropriate controls to eliminate order effects.

Outcome measures

We will examine the effects of reward and TBS and their interaction on measures of learning. Secondary outcome measures will be how TBS and reward interact to alter the pattern of BOLD activation on MRI and the effects of relevant genetic variation on learning variables and BOLD activation. We will examine the effects of genetic variations in relevant genes on these outcomes.

ELIGIBILITY:
* Participants will be 272 healthy volunteers drawn from the population in the NIH clinical research volunteer program.

INCLUSION CRITERIA:

Healthy

Right-handed

Ages 18-70 (inclusive)

Have completed high school or college in an English speaking country.

All participants must have had a neurological examination by a NINDS physician within the last two years.

All participants in the fMRI experiments must also have had a clinical MRI within the last year.

EXCLUSION CRITERIA:

Individuals with conditions that could pose a risk relating to the safety of the MRI procedure will be excluded from the protocol such as:

Those with ferromagnetic metal in the cranial cavity or eye, e.g. aneurysm clip, implanted neural stimulator, cochlear implant, ocular foreign body.

Those with an implanted cardiac pacemaker or auto-defibrillator.

Those with an insulin pump.

Those with an irremovable body piercing.

Pregnant women

Individuals with conditions that could pose a risk relating to the safety of the TMS procedure will be excluded from the protocol such as:

* Those with significant abnormality on neurological examination.
* Those with metal in the cranial cavity or eye, e.g. aneurysm clip, implanted neural stimulator, cochlear implant, ocular foreign body.
* Those with an implanted cardiac pacemaker or auto-defibrillator.
* Those with an insulin pump.
* Pregnant women

Individuals with conditions that could compromise our interpretation of the TBS and fMRI results will be excluded such as:

* Those with significant abnormality on neurological examination.
* Those who have a significant psychiatric illness or have a history of psychiatric illness.
* Those using medication affecting the DA system, such as phenothiazine antihistamines (promethazine), antiemetics or decongestants within the last month.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-12-07; Study Completion 2017-06-23

PRIMARY OUTCOMES:
We will examine the effects of reward and TBS and their interaction on measures of learning. | One hour

SECONDARY OUTCOMES:
Secondary outcome measures will be how TBS and reward interact to alter the pattern of BOLD activation on MRI and the effects of relevant genetic variation on learning variables and BOLD activation. | One hour

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arancio O, Chao MV. Neurotrophins, synaptic plasticity and dementia. Curr Opin Neurobiol. 2007 Jun;17(3):325-30. doi: 10.1016/j.conb.2007.03.013. Epub 2007 Apr 6. PMID 17419049
- [Background] Aron AR, Gluck MA, Poldrack RA. Long-term test-retest reliability of functional MRI in a classification learning task. Neuroimage. 2006 Feb 1;29(3):1000-6. doi: 10.1016/j.neuroimage.2005.08.010. Epub 2005 Sep 1. PMID 16139527
- [Background] Badgaiyan RD, Fischman AJ, Alpert NM. Striatal dopamine release in sequential learning. Neuroimage. 2007 Nov 15;38(3):549-56. doi: 10.1016/j.neuroimage.2007.07.052. Epub 2007 Aug 15. PMID 17888684